CLINICAL TRIAL: NCT00305019
Title: A Double- Blind, Randomized, Placebo-Controlled Study to Evaluate the Safety and Antiviral Activity of Clevudine 30 Mg QD and 50 Mg QD Doses in Patients Infected With Hepatitis B Virus
Brief Title: Safety and Antiviral Activity of Clevudine in Patients Infected With Hepatitis B Virus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bukwang Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L-FMAU-201
Record Dates: First submitted 2006-03-17; First posted 2006-03-21 (Estimated); Last update posted 2006-04-12 (Estimated); Status verified 2006-04

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — clevudine

INTERVENTIONS:
Drug: clevudine

SUMMARY:
The purpose of this study is to determine the antiviral effects and safety of clevudine 30 mg once a day (QD) and 50 mg QD in patients infected with hepatitis B virus (HBV).

ELIGIBILITY:
Inclusion Criteria:

1. Patient who is between 18 and 60 years of age, inclusive
2. Patient who is HBV DNA positive with DNA levels at screening more than 3 x 10^6 copies/mL.
3. Patient who is documented to be hepatitis B surface antigen (HBsAg) positive for > 6 months. Patient is HBeAg positive and anti-HBe negative.

   Evidence of HBsAg (+) for the previous 6 months may include the following:
   * documentation of HBsAg (+) for the previous 6 months
   * documentation of HBsAg (+) for the previous 3 months and IgM anti-HBc negative at screening
   * IgM anti-HBc negative and IgG anti-HBc positive at screening
4. Patient who has ALT levels which are in the range of more than 2 to less than 10 times the upper limit of normal (x ULN) and bilirubin levels < 1.5 x ULN.
5. Female patient with a negative serum (HCG) pregnancy test taken within 14 days of starting therapy.
6. Patient who is able to give written informed consent prior to study start and to comply with the study requirements.
7. Patients who continue to meet the following criteria after completion of the Week 36 visit will have additional follow-up visits at Week 40, 44, 48:

   * have received no additional therapy since completion of 12 weeks of treatment of L-FMAU and
   * continue with period 1 log10 decrease in HBV DNA from baseline.

Exclusion Criteria:

1. Patient who is currently receiving antiviral, immunomodulatory or corticosteroid therapy.
2. Patients previously treated with lamivudine, lobucavir, adefovir or any other investigational nucleoside for HBV infection.
3. Patients with previous treatment with interferon that have ended less than 6 months prior to the screening visit.
4. Patient who has a history of ascites, variceal hemorrhage or hepatic encephalopathy.
5. Patient who is coinfected with hepatitis C virus (HCV), hepatitis D virus (HDV) or HIV.
6. Patient with clinical evidence of cirrhosis or hepatocellular carcinoma
7. Patient who is pregnant or breast-feeding.
8. Patient who is unwilling to use an "effective" method of contraception during the study and for up to 30 days after the use of study drug ceases. For males, condoms should be used. Females must be surgically sterile (via hysterectomy or bilateral tubal ligation), post-menopausal or using at least a medically acceptable barrier method of contraception (i.e., intrauterine device [IUD], barrier methods with spermicide or abstinence)
9. Patient who has a clinically relevant history of abuse of alcohol or drugs.
10. Patient who has a significant gastrointestinal, renal, hepatic (decompensated), bronchopulmonary, neurological, cardiovascular, oncologic or allergic disease.
11. Patient who has creatinine clearance less than 60 mL/min as estimated by the following formula:

(140-age in years) (body weight [kg])/ (72) (serum creatinine [mg/dL]) [Note: multiply estimates by 0.85 for women]

Patients found to have tyrosine, methionine, aspartate, aspartate (YMDD) HBV DNA polymerase mutation after the enrollment will be excluded from the efficacy evaluation but included in the safety evaluation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120
Dates: Start 2002-07; Study Completion 2004-03

PRIMARY OUTCOMES:
Efficacy: Change from baseline in HBV DNA (log10)

SECONDARY OUTCOMES:
Efficacy: Proportion of patients with HBV DNA below 1 pg/mL
Proportion of patients with HBV DNA below the assay limit of detection (LOD) (SuperDigene HC test II LOD, <4,700 copies/mL)
Proportion of patients with hepatitis Be antigen (HBeAg) loss
Seroconversion rate (HBeAg loss and hepatitis Be antibody [HBeAb] positivity)
Biochemical improvement (e.g., ALT normalization)
Safety
Laboratory tests
Adverse Events
Vital Signs
Electrocardiogram (ECG)

CONTACTS AND LOCATIONS:
Overall Officials: Hyo Suk Lee, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (8):
- South Korea (8):
  - Korea University Guro Hospital, Guro-dong, Guro-ku, Seoul
  - Seoul National University, Yeongeon-dong, Jongno-Gu, Seoul
  - Kangdong Sacred Heart Hospital, Gildong, Kangdong-Gu, Seoul
  - Samsung Medical Center, Ilwon-dong, Kangnam-Gu, Seoul
  - Yongdong Severance Hospital, Togok-tong, Kangnam-Gu, Seoul
  - Asan Medical Center, P’ungnabi-dong, Songpa-Gu, Seoul
  - Ewha Womans University Hospital, Mokdong, Yangchon-Gu, Seoul
  - St. Mary's Hospital, Youido, Yougdungpo-Gu, Seoul

REFERENCES:
- [Derived] Lee HS, Chung YH, Lee K, Byun KS, Paik SW, Han JY, Yoo K, Yoo HW, Lee JH, Yoo BC. A 12-week clevudine therapy showed potent and durable antiviral activity in HBeAg-positive chronic hepatitis B. Hepatology. 2006 May;43(5):982-8. doi: 10.1002/hep.21166. PMID 16628625